CLINICAL TRIAL: NCT01408654
Title: Social Connections and Healthy Aging (The Senior Connection)
Acronym: TSC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Yeates Conwell, Co-Chair, Department of Psychiatry, Professor of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1U01CE001942-01 (NIH)
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Suicidal Ideation; Depression
Keywords: Suicidal Ideation; Loneliness; Social Support; Voluntary Workers; Friends/Companions; Prevention; Aged
MeSH Terms: conditions — Suicidal Ideation; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peer Companionship (Experimental): Behavioral intervention: Receipt of peer companionship provided by trained, supervised volunteer companions.
  Interventions: Behavioral: Peer Companionship
- Care-as-Usual (No Intervention): Care-as-Usual in Primary Care

INTERVENTIONS:
Behavioral: Peer Companionship — Peer companionship is provided at least four times per month over two years in the form of friendly visiting, supportive phone calls, and some instrumental support.
  Other Names: Intervention is administered to the peer companionship arm.
  Arms: Peer Companionship

SUMMARY:
This randomized trial compares peer companionship to care-as-usual in primary care on the outcome of risk for suicidal behavior in late life. The investigators hypothesize that older adults assigned to receive peer companionship will report greater social connectedness and less death and suicidal ideation compared to older adults assigned to care as usual.

DETAILED DESCRIPTION:
There is a pressing need for interventions that reduce risk for suicide in later life. Older adults in the U.S. have the highest rate of suicide and are the fastest growing segment of the population. The investigators can anticipate a large rise in the number of older adults who die by suicide in coming decades. This application is in response to RFA-CE-10-006. Consistent with the CDC's key strategy of reducing suicide by promoting connectedness, our long-term goal is to reduce late life suicide-related morbidity and mortality by leveraging the resources and expertise of the aging services provider network (ASPN) to address unmet social needs of community-dwelling older adults. Our objectives with this proposal are (1) to examine whether linking socially disconnected seniors with peer supports through the Retired and Senior Volunteer Program (RSVP) is effective in reducing risk for suicide, and (2) to test an hypothesized mechanism for the association of social disconnectedness and suicidal ideation and behavior informed by the Interpersonal Theory of Suicide.

The investigators will recruit 400 primary care patients (200 men and 200 women) over age 60 years who endorse feeling lonely and/or as if they are a burden on others. They will be randomly assigned to either of two conditions. Those assigned to The Senior Connection (TSC) will either be paired with a peer companion or, if they prefer and are eligible, be trained and placed as a peer companion for others by RSVP. The comparison group will receive no further intervention ("care-as-usual" [CAU]). Subjects will be followed for up to 24 months with repeated in-home (baseline, 12, and 24 months) and telephone assessments (3, 6, and 18 months).

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older
* Primary Care Patient
* Endorses feeling lonely and/or like a burden in the the past two weeks

Exclusion Criteria:

* Positive dementia screen
* Current alcohol abuse
* Psychosis
* Suicidal ideation with intent to act (current or past month.)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2011-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Suicidal Ideation | Baseline, 3,6,12,18,24 months
  Severity of suicidal and death ideation assessed with the Geriatric Suicide Ideation Scale

SECONDARY OUTCOMES:
Social Connectedness | Baseline, 3,6,12,18,24 months
  Thwarted belongingness and perceived burdensomeness assessed by the Interpersonal Needs Questionnaire.
Connectedness | Baseline, 3,6,12,18,24 months
  Social network size/density/quality assessed with the National Social Life, Health, and Aging Project Social Network Module.
Depression | Baseline, 3,6,12,18,24 months
  Assessed with the PHQ-9

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester School of Medicine and Dentistry, Rochester, New York, United States

REFERENCES:
- [Background] Van Orden KA, Stone DM, Rowe J, McIntosh WL, Podgorski C, Conwell Y. The Senior Connection: design and rationale of a randomized trial of peer companionship to reduce suicide risk in later life. Contemp Clin Trials. 2013 May;35(1):117-26. doi: 10.1016/j.cct.2013.03.003. Epub 2013 Mar 16. PMID 23506973
- [Derived] Parkhurst KA, Daks JS, Conwell Y, Podgorski CA, Van Orden KA. Social network subtypes among socially disconnected older adults at risk for suicide: A latent class analysis. Suicide Life Threat Behav. 2022 Oct;52(5):963-974. doi: 10.1111/sltb.12893. Epub 2022 Jun 23. PMID 35735167